CLINICAL TRIAL: NCT01912625
Title: A Phase 1 Study of Trametinib in Combination With Chemoradiation for KRAS Mutant Non-small Cell Lung Cancer
Brief Title: Trametinib, Combination Chemotherapy, and Radiation Therapy in Treating Patients With Stage III Non-small Cell Lung Cancer That Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01357; NCI-2013-01357 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-1053; 763093; 9448 (Other: M D Anderson Cancer Center); 9448 (Other: CTEP); P30CA016672 (NIH); P50CA070907 (NIH); U01CA062461 (NIH); UM1CA186688 (NIH); UM1CA186712 (NIH)
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Recurrent Lung Non-Small Cell Carcinoma; Stage III Lung Non-Small Cell Cancer AJCC v7; Stage IIIA Lung Non-Small Cell Cancer AJCC v7; Stage IIIB Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy, Conformal; Carboplatin; Radiotherapy, Image-Guided; Radiotherapy, Intensity-Modulated; Paclitaxel; Taxes; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (trametinib, chemotherapy, radiation therapy) (Experimental): CONCURRENT CHEMOTHERAPY: Patients undergo IMRT or 3D-CRT QD 5 days a week for 6 weeks. Patients receive trametinib PO QD and carboplatin IV over 30 minutes and paclitaxel IV over 1 hour once weekly. Treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients without disease progression after completion of chemoradiation proceed to consolidation chemotherapy.
  CONSOLIDATION CHEMOTHERAPY: Beginning 3 weeks after completion of concurrent chemoradiation, patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on days 1 and 22. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Carboplatin; Radiation: Image Guided Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Pharmacological Study; Drug: Trametinib

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D-CRT
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D radiotherapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal; Three dimensional external beam radiation therapy (procedure)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Radiation: Image Guided Radiation Therapy — Undergo IGRT
  Other Names: IGRT; image-guided radiation therapy; Image-Guided Radiotherapy
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Pharmacological Study — Correlative studies
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212

SUMMARY:
This phase I trial studies the side effects and the best dose of trametinib when given together with combination chemotherapy and radiation therapy in treating patients with stage III non-small cell lung cancer that cannot be removed by surgery. Trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells. Giving trametinib, combination chemotherapy, and radiation therapy may be a better treatment for non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum-tolerated dose (MTD) of GSK1120212 (trametinib) combined with standard chemoradiation in unresectable non-small cell lung cancer (NSCLC) and safety as measured by the rate of grade 3 or worse non-hematological toxicities occurring prior to the beginning of consolidation therapy (including all toxicities attributed to chemoradiation occurring within 10 weeks of the start of radiation therapy).

II. Pharmacokinetic (PK) analysis of carboplatin, paclitaxel, and trametinib.

SECONDARY OBJECTIVES:

I. Response rate based on computed tomography (CT) or fludeoxyglucose F 18 (FDG)-positron emission tomography (PET)/CT imaging response assessment after completion of chemoradiation.

II. Biomarker correlate to response and resistance. III. Overall survival. IV. Patterns of recurrence. V. Determine dose delay and the percentage of dose delivered for each agent.

OUTLINE: This is a dose-escalation study of trametinib.

CONCURRENT CHEMOTHERAPY: Patients undergo intensity-modulated radiation therapy (IMRT) or three-dimensional conformal radiotherapy (3D-CRT) once daily (QD) 5 days a week for 6 weeks. Patients receive trametinib orally (PO) QD and carboplatin intravenously (IV) over 30 minutes and paclitaxel IV over 1 hour once weekly. Treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients without disease progression after completion of chemoradiation proceed to consolidation chemotherapy.

CONSOLIDATION CHEMOTHERAPY: Beginning 3 weeks after completion of concurrent chemoradiation, patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on days 1 and 22. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed, newly diagnosed or recurrent from a previously treated early stage lung cancers that are locally confined, non-small cell lung cancers that are considered unresectable and for which chemoradiation will be considered definitive therapy; patients with recurrent cancer that is amendable for chemoradiation can be eligible only if patients with prior lobectomy for stage I cancer had not had adjuvant chemotherapy, and more than 8 weeks have elapsed from surgery to allow for wound healing; patients who recur from prior X-ray therapy (XRT) or stereotactic body radiation therapy (SBRT) will not be eligible
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Prior thoracic radiation allowed only if there is minimal to no overlap with the treatment area estimated at the time of consultation, and there is no cumulative esophageal dose that exceeds more than 50% of the maximal acceptable dose tolerance
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Life expectancy of greater than 6 months
* Able to swallow and retain orally-administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Hemoglobin >= 9 g/dL
* Platelets >= 100 x 10^9/L
* Albumin >= 2.5 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional ULN
* Serum creatinine =< 1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) >= 50 mL/min OR 24-hour urine creatinine clearance >= 50 mL/min
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 x institutional ULN
* Left ventricular ejection fraction >= institutional lower limit of normal (LLN) by echocardiogram (ECHO) or multi gated acquisition scan (MUGA)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the study participation, and for four months after the last dose of the drug; women of child-bearing potential must have a negative serum pregnancy test within 14 days prior to registration and agree to use effective contraception throughout the treatment period and for 4 months after the last dose of study treatment; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Activating Kirsten rat sarcoma viral oncogene homolog (KRAS) mutation (any G12, G13, Q61) confirmed by Clinical Laboratory Improvement Act (CLIA)-certified testing
* The availability of formalin-fixed paraffin embedded archival tissue from core biopsy of tumors is recommended for exploratory analysis

Exclusion Criteria:

* History of another malignancy

  * Exception: patients who have been disease-free for 3 years, or patients with a history of completely resected non-melanoma skin cancer and/or patients with indolent secondary malignancies, are eligible; consult the Cancer Therapy Evaluation Program (CTEP) Medical Monitor if unsure whether second malignancies meet the requirements specified above
* History of interstitial lung disease or pneumonitis
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 21 days prior to enrollment
* Use of other investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of trametinib and during the study
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trametinib, or excipients or to dimethyl sulfoxide (DMSO) or to either carboplatin or paclitaxel
* Current use of a prohibited medication; the following medications or non-drug therapies are prohibited:

  * Other anti-cancer therapy while on study treatment; (note: megestrol [Megace] if used as an appetite stimulant is allowed)
  * Concurrent treatment with bisphosphonates is permitted; however, treatment must be initiated prior to the first dose of study therapy; prophylactic use of bisphosphonates in patients without bone disease is not permitted, except for the treatment of osteoporosis
  * Concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, St. John's wort, kava, ephedra [ma huang], gingko biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, or ginseng)
* History or current evidence/risk of retinal vein occlusion (RVO)
* History or evidence of cardiovascular risk including any of the following:

  * Left ventricular ejection fraction (LVEF) < LLN
  * A QT interval corrected for heart rate using the Bazett's formula corrected QT (QTcB) >= 480 msec
  * History or evidence of current clinically significant uncontrolled arrhythmias (exception: patients with controlled atrial fibrillation for > 30 days prior to registration are eligible)
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to registration
  * History or evidence of current >= class II congestive heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
  * Known cardiac metastases
* Known hepatitis B virus (HBV), or hepatitis C virus (HCV) infection (patients with chronic or cleared HBV and HCV infection are eligible); patients with human immunodeficiency virus (HIV) are not eligible if on anti-retroviral medications
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women or nursing mothers; women of childbearing potential should be advised to avoid pregnancy and use effective methods of contraception; men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception; if a female patient or a female partner of a patient becomes pregnant while the patient receives trametinib, the potential hazard to the fetus should be explained to the patient and partner (as applicable)
* HIV-positive patients on combination antiretroviral therapy are ineligible
* Patients who do not consent for PK studies to be performed (alternatively: patients who initially consent to be on study but withdraws consent for PK study will be taken off study and replaced)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-10-28 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity defined as any grade 3 or 4 non-hematologic toxicities according to Common Terminology Criteria for Adverse Events version 4.0 grading | Within 70 days from the start of radiation therapy
  Toxicity will be tabulated by dose, type, and grade. The probability of toxicity over 70 days as a function of dose will be estimated by fitting a Bayesian binary outcome regression model.
Pharmacokinetic parameters of carboplatin and paclitaxel with the dosing of trametinib | At 15 and 30 minutes prior to the start of infusion and then at 30 minutes, 4, 10, and 24 hours after infusion on day 15

SECONDARY OUTCOMES:
Response rate based on CT or FDG-PET/CT imaging response assessment after completion of chemoradiation | Up to 4 years
  Response rate will be estimated and 95% confidence interval will be provided.
Overall survival (OS) | Up to 4 years
  Unadjusted OS will be estimated by the Kaplan and Meier method.
Patterns of recurrence | Up to 4 years
  Relapse-free survival will be estimated by the Kaplan and Meier method.
KRAS mutation status | Baseline
  KRAS and other biomarkers will be compared between pre-treatment tumors and recurrent tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Lin, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - M D Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin